CLINICAL TRIAL: NCT02502331
Title: A Randomized, Observer Blinded, Controlled Trial to Evaluate the Safety and Immunogenicity of a New Formulation of Euvichol® (Killed Bivalent Whole Cell Oral Cholera Vaccine Manufactured by EuBiologics Co. Ltd.) in Healthy Individuals
Brief Title: Safety and Immunogenicity of a New Formulation of Euvichol®
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Vaccine Institute (Other)
Collaborators: EuBiologics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IVI-CHOVI-EUVICHOL
Record Dates: First submitted 2015-07-14; First posted 2015-07-20 (Estimated); Last update posted 2015-12-17 (Estimated); Status verified 2015-12

CONDITIONS: Cholera
Keywords: Oral Cholera Vaccine; immunogenicity; safety
MeSH Terms: conditions — Cholera

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- study group (Experimental): Test Oral Cholera Vaccine
  Interventions: Biological: Test Oral Cholera Vaccine
- comparator group (Active Comparator): Euvichol®
  Interventions: Biological: Euvichol®

INTERVENTIONS:
Biological: Test Oral Cholera Vaccine — Thimerosal free, manufactured at 600 L scale killed bivalent (O1 and O139) whole cell-oral cholera vaccine (WC-OCV) manufactured by Eubiologics Co., Ltd.
  Arms: study group
Biological: Euvichol® — Licensed, manufactured at 100 L scale killed bivalent (O1 and O139) whole cell-oral cholera vaccine (WC-OCV) manufactured by Eubiologics Co., Ltd.
  Arms: comparator group

SUMMARY:
* Number of doses and intervals: Two doses, 2 weeks apart
* Method of administration: Oral administration
* Volume of vaccine to be administered: 1.5 mL/dose
* Observational period: 4 weeks (2 weeks after each dose)
* Number of visits: 3 visits

  1. Visit 1: Screening and enrollment (1st dosing)
  2. Visit 2: 2nd dosing 2 weeks after 1st dose (14+3 days)
  3. Visit 3: 2 weeks after the 2nd dose (28+3 days), end of subject participation. This study will be carried out in healthy adults and children, at two sites, enrollment will be competitive between the sites. Subjects will be stratified according to age into adults (18~40 years of age) and children (1~17 years of age). According to the pre-generated randomization list, the participants will be randomized to the test or comparator groups (Visit 1) and will be given either the test vaccine or the comparator vaccine. For immunogenicity assessment, blood sample will be taken at Visit 1 (prior to vaccination), Visit 2 (prior to vaccination), and at the end-of-study Visit (Visit 3). For Safety assessment: the participants will be observed for 30 minutes post vaccination and instructed to record solicited adverse events that occur up to 6 days after vaccination on the participant diary card.

This study is observer-blind: vaccine administrator and vaccine safety evaluator will be two distinct persons to avoid bias of safety assessment. Trial staff other than the vaccine administrator will remain blinded and will not handle the investigational product.

DETAILED DESCRIPTION:
1. Primary immunogenicity endpoint

   * Geometric Mean Titer (GMT) of Vibriocidal antibodies against Inaba serogroup O1 post second dose
   * GMTof Vibriocidal antibodies against Ogawa serogroup O1 post second dose
   * GMT of Vibriocidal antibodies against serogroup O139 post second dose
2. Secondary immunogenicity endpoints

   * Proportion of participants showing seroconversion against Inaba serogroup O1, Ogawa serogroup O1and serogroup O139 post vaccinations
   * Seroconversion is defined as 4-fold rise in vibriocidal antibody titer at Visit 3 two weeks after the second dose, compared to baseline titers, measured at Visit 1 prior to vaccination.

Proportion of participants with:

1. Immediate reactions within 30 minutes after each dose of vaccination.
2. Solicited systemic Adverse Events: nausea/vomiting, diarrhea, headache, fatigue, myalgia, fever, and anorexia/loss of appetite within 7 days after each vaccination.

   1. Diarrhea is defined as having 3 or more loose/watery stools within a 24-hour period or at least 1 bloody loose stool or any number of loose stools with signs of dehydration.
   2. Fever is defined as having an axillary temperature of 38 ℃
3. Unsolicited Adverse Events and Serious Adverse Events occurring 14 days following each vaccination, as reported by participants Measurement of Geometric Mean Titer of vibriocidal antibodies post vaccination, Ratio ofGeometric Mean Titer of vibriocidal antibodies post vaccination of Test vaccine' compared with 'Comparator vaccine'.

Expected outcome: Statistical equivalence of the two vaccines.

ELIGIBILITY:
Inclusion Criteria:

1. Subject willing to provide written informed consent to study participation voluntarily provided by an individual or his/her legally acceptable representative.
2. Individuals aged 1 - 40 years.
3. An individual who can be followed up during the study period and is capable of complying with the study requirements

Exclusion Criteria:

1. Known history of hypersensitivity reactions to other preventive vaccines.
2. Known history of immune function disorders including immunodeficiency diseases, or chronic use of systemic steroids (> 20 mg/day prednisone equivalent for periods exceeding 10 days), cytotoxic drugs or other immunosuppressants.
3. Severe chronic diseases, based on the judgment of the investigator.
4. 38℃ or higher body temperature measured prior to investigational product dosing.
5. Abdominal pain, nausea, vomiting, or decreased appetite within 24 hours prior to study initiation.
6. Diarrhea or administration of antidiarrheal drugs or antibiotics to treat diarrhoea within 1 week prior to study initiation.
7. Diarrhea or abdominal pain lasting 2 weeks or longer within 6 months prior to study initiation.
8. Other vaccination within 1 week prior to study initiation or planned vaccination during the study, except for tetanus toxoid vaccine.
9. Participation in another clinical trial with investigational product dosing within 1 month prior to study initiation.
10. Pregnant or lactating women, women of reproductive age planning pregnancy and/or lactation before the end of the study period.
11. An individual thought to have difficulty participating in the study due to other reasons, based on the judgment of the investigator
12. History of cholera vaccinations or history of cholera.
13. History of alcohol or substance abuse
14. Participant planning to move from the study area before the end of study period.

Ages: 1 Year to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 442 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-06 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Immunogenicity endpoint for Inaba O1 | 28 days
  Geometric Mean Titer (GMT) of Vibriocidal antibodies against Inaba serogroup O1 post second dose
Immunogenicity endpoint for Ogawa O1 | 28 days
  GMTof Vibriocidal antibodies against Ogawa serogroup O1 post second dose
Immunogenicity endpoint O139 | 28 days
  GMT of Vibriocidal antibodies against serogroup O139 post second dose

SECONDARY OUTCOMES:
Proportion of participants showing seroconversion against Inaba serogroup O1, Ogawa serogroup O1and serogroup O139 post vaccinations. | 28 days
Seroconversion is defined as 4-fold rise in vibriocidal antibody titer at Visit 3 two weeks after the second dose, compared to baseline titers, measured at Visit 1 prior to vaccination. | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Laura Digilio, MD, Principal Investigator — International Vaccince Institute

REFERENCES:
- [Derived] Russo P, Ligsay AD, Olveda R, Choi SK, Kim DR, Park JY, Park JY, Syed KA, Dey A, Kim YH, Lee SH, Kim J, Chon Y, Digilio L, Kim CW, Excler JL. A randomized, observer-blinded, equivalence trial comparing two variations of Euvichol(R), a bivalent killed whole-cell oral cholera vaccine, in healthy adults and children in the Philippines. Vaccine. 2018 Jul 5;36(29):4317-4324. doi: 10.1016/j.vaccine.2018.05.102. Epub 2018 Jun 9. PMID 29895500